CLINICAL TRIAL: NCT02268344
Title: Brief Intraoperative Electrical Stimulation for Prevention of Shoulder Dysfunction After Oncologic Neck Dissection (ESSAN): a Double-blinded, Randomized Control Trial
Brief Title: Brief Intraoperative Electrical Stimulation for Prevention of Shoulder Dysfunction After Oncologic Neck Dissection
Acronym: ESSAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: pro00046671
Record Dates: First submitted 2014-10-10; First posted 2014-10-20 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Shoulder Pain; Head Neck Cancer
Keywords: nerve regeneration; spinal accessory nerve; shoulder function; head neck cancer; electrical stimulation
MeSH Terms: conditions — Shoulder Pain; Head and Neck Neoplasms | interventions — Electric Stimulation

STUDY DESIGN:
Intervention Model Description: Brief intraoperative electrical stimulation of the spinal accessory nerve (ESSAN) continuously at 20 Hz, 10-15V for 60 minutes immediately following neck dissection
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Grass SD9 Stimulator (Active Comparator): Brief intraoperative electrical stimulation of the spinal accessory nerve (ESSAN) continuously at 20 Hz, 10-15V for 60 minutes immediately following neck dissection.
  Interventions: Device: Grass SD9 Stimulator
- No Stimulation (No Intervention): No stimulation will be performed in this group, and patients will simply have the neck dissection as planned. No sham stimulation is required, as all outcome measures are performed by individuals not present in the operating room, and therefore, blinded to the treatment arm.

INTERVENTIONS:
Device: Grass SD9 Stimulator — Electrical stimulation will be applied to the nerve using the Grass SD9 Stimulator at a frequency of 20Hz, 10-15V, for 60 minutes during the surgery. This will occur after the neck dissection has been completed, and the remainder of the surgery will continue during stimulation. The stimulation will be applied using the Grass SD9 Stimulator and the current will be conducted to the nerve using a sterile wire electrode that will be encircled around the nerve at its most proximally-exposed portion (skull base). The wire will be removed after 60 minutes of stimulation has been applied.
  Other Names: Electrical Stimulation (ES)
  Arms: Grass SD9 Stimulator

SUMMARY:
Introduction: Shoulder pain and dysfunction is common after oncologic neck dissection for head and neck cancer (HNC). These symptoms can hinder postoperative rehabilitation and oral hygiene, activities of daily living (ADLs), and return to work after treatment. Due to the rising incidence of Human papillomavirus (HPV)-associated oropharyngeal cancer, patients are often diagnosed in the 3rd or 4th decade of life, leaving many potential working years lost. Brief electrical stimulation (BES) is a novel technique that has been shown to enhance neuronal regeneration after injury through a brain-derived neurotrophic growth factor (BDNF)-driven molecular pathway. The aim of this study is to examine the utility of intraoperative BES in prevention of shoulder pain and dysfunction after oncologic neck dissection.

Methods: All adult patients with a new diagnosis of HNC undergoing surgery with neck dissection including Level IIb and postoperative radiotherapy will be enrolled. Patients will undergo intraoperative BES after completion of neck dissection for 60 minutes continuously at 20 Hz with an intensity of 1.5 times the motor threshold. Postoperatively, patients will be evaluated using the Constant-Murley Shoulder Score, a scale that assesses shoulder pain, activities of daily living (ADLs), strength, and range of motion. Secondary outcomes measured will include scores on the Oxford Shoulder Score, the Neck Dissection Impairment Index (NDII), and the University of Washington Quality of Life (UW-QOL) score. Primary and secondary outcomes will be assessed at 1, 2, 3, 6, and 12 months postoperatively. Study and placebo groups will be compared using a Mann-Whitney analysis.

DETAILED DESCRIPTION:
This study will be conducted as a randomized, double-blinded, placebo-controlled trial. Two parallel treatment groups will be examined with a 1:1 allocation: 1) brief intraoperative electrical stimulation continuously at 20 Hz at an intensity of 1.5 times the motor threshold for 60 minutes, or 2) sham/no stimulation for 60 minutes. Individuals will be allocated to treatment groups using a block randomization sequence. Participants and researchers measuring outcomes will be blinded to treatment groups. Stimulation (BES or sham) will occur intraoperatively immediately following neck dissection for 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years
* New adult head and neck cancer patients
* Undergoing major resection and reconstruction surgery including oncologic neck dissection including Level IIb
* Undergoing adjuvant therapy

Exclusion Criteria:

* Oncologic resection necessitating unilateral or bilateral resection of the sternocleidomastoid, SAN, partial resection of trapezius muscle, hypoglossal nerve, skin, carotid resection, or deep muscle resection
* Previous surgery or radiation therapy to the head and/or neck
* Recurrent head and neck cancer
* Preoperative, pre-existing shoulder dysfunction or weakness, including myopathy, neuropathy, or arthropathy
* Presence of existing implanted electrical device (eg. pacemaker, deep brain stimulator, vagal nerve stimulator
* Previous or current neurological disease which may adversely affect shoulder dysfunction
* Unable to read, write, and speak English
* Lacking capacity to give consent
* Unwilling to present for follow-up appointments or follow-up objective shoulder assessment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2014-10-06 (Actual); Primary Completion 2015-06-06 (Actual); Study Completion 2015-06-06 (Actual)

PRIMARY OUTCOMES:
Constant-Murley Score | 6 months postoperatively
  The Constant-Murley score is a 100-point scale composed of a number of individual parameters, detailing the level of shoulder pain and the ability to carry out normal daily activities of the patient. The Constant-Murley Score is a 100-point scale composed of a number of individual parameters, designed to determine functionality after shoulder treatment. It includes includes 4 subscales that assess pain, activities of daily living, strength, and range of motion (forward elevation, external rotation, abduction, and internal rotation of the shoulder). A higher score indicates higher quality of function.

SECONDARY OUTCOMES:
Oxford Shoulder Score (OSS) | 6 months postoperatively
  The OSS is a 12-item, multi-dimensional, self-report questionnaire regarding shoulder-specific daily activity in the previous 4 weeks.
Neck Dissection Impairment Index (NDII) | 6 months postoperatively
  The Neck Dissection Impairment Index (NDII), is a 10-item self-report questionnaire using a 5-point Likert scale for assessment of shoulder impairment after neck dissection.
Nerve Conduction Studies (NCS) | 6 months months postoperatively
  This will include conduction velocity and amplitude as it relates to nerve injury during oncologic neck dissection.
Electromyographic (EMG) studies | 6 months postoperatively
  This will pertain to electrophysiologic thresholds necessary to evoke a motor response from the trapezius and sternocleidomastoid, to evaluate nerve function.
University of Washington Quality of Life (UW-QOL) questionnaire | 6 months postoperatively
  This instrument will be used to asses quality of life (QOL) differences between the study and placebo groups following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Brittany Barber, MD, Study Chair — Division of Otolaryngology-Head & Neck Surgery, University of Alberta; Daniel O'Connell, MD MSc FRCSC, Principal Investigator — Division of Otolaryngology-Head & Neck Surgery, University of Alberta; Hadi Seikaly, MD MAL FRCSC, Study Director — Division of Otolaryngology-Head & Neck Surgery, University of Alberta; Ming Chan, MD FRCPC, Study Director — Department of Physical Rehabilitation and Medicine, University of Alberta; Margaret McNeely, PT PhD, Study Director — Faculty of Rehabilitation Medicine, University of Alberta; Jeffrey Harris, MD MHA FRCSC, Study Chair — Division of Otolaryngology-Head & Neck Surgery, University of Alberta; Jaret Olson, MD FRCSC, Study Chair — Division of Plastic Surgery, University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Barber B, Seikaly H, Ming Chan K, Beaudry R, Rychlik S, Olson J, Curran M, Dziegielewski P, Biron V, Harris J, McNeely M, O'Connell D. Intraoperative Brief Electrical Stimulation of the Spinal Accessory Nerve (BEST SPIN) for prevention of shoulder dysfunction after oncologic neck dissection: a double-blinded, randomized controlled trial. J Otolaryngol Head Neck Surg. 2018 Jan 23;47(1):7. doi: 10.1186/s40463-017-0244-9. PMID 29361981
- [Derived] Barber B, McNeely M, Chan KM, Beaudry R, Olson J, Harris J, Seikaly H, O'Connell D. Intraoperative brief electrical stimulation (BES) for prevention of shoulder dysfunction after oncologic neck dissection: study protocol for a randomized controlled trial. Trials. 2015 May 30;16:240. doi: 10.1186/s13063-015-0745-7. PMID 26021563